CLINICAL TRIAL: NCT04580914
Title: Clinical Evaluation of the StablePoint Catheter and Force Sensing System for Paroxysmal Atrial Fibrillation
Acronym: NEwTON AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92567361
Record Dates: First submitted 2020-09-21; First posted 2020-10-09 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation; StablePoint; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment with Ablation Catheter (Experimental): Patients who undergo treatment with the ablation catheter for the treatment of paroxysmal atrial fibrillation
  Interventions: Device: Treatment with IntellaNav StablePoint Ablation Catheter

INTERVENTIONS:
Device: Treatment with IntellaNav StablePoint Ablation Catheter — Patients will be treated with an ablation catheter
  Other Names: IntellaNav StablePoint Catheter System

SUMMARY:
The NEwTON AF study is a multi-center, global, prospective, single arm study to establish the safety and effectiveness of the IntellaNav StablePoint Catheter and Force-Sensing System in subjects with symptomatic, drug refractory, recurrent paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. History of recurrent symptomatic Paroxysmal Atrial Fibrillation (PAF), defined as atrial fibrillation (AF) that terminates spontaneously or with intervention (either procedure or drug therapy) within seven days of onset. Minimum documentation includes the following:

   a physician's note indicating recurrent self-terminating atrial fibrillation (AF) which includes at least two symptomatic AF episodes in the patient's history within the last 6 months prior to enrollment, and any electrocardiographically documented AF episode within 12 months prior to enrollment.
2. Subjects who are eligible for an ablation procedure for PAF according to 2017 HRS expert consensus statement on catheter ablation of atrial fibrillation;
3. Subjects refractory or intolerant to at least one class I or class III antiarrhythmic medication or contraindicated to any class I or class III medications;
4. Subjects who are willing and capable of providing informed consent;
5. Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center;
6. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Subjects with New York Heart Association (NYHA) Class III or IV heart failure < 180 days prior to enrollment
2. Left atrial diameter > 5.0 cm or left atrial volume >50 ml/m² indexed based on the most recent echocardiography+
3. Left ventricular ejection fraction < 35% based on the most recent echocardiogram +
4. Continuous AF lasting longer than seven (7) days
5. Subjects who have undergone any previous left atrial cardiac ablation (RF, Cryo, surgical)
6. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
7. Subjects who have undergone any cardiac ablation or any surgery within 30 days prior to enrollment
8. Currently implanted with a pacemaker, ICD, CRT device, or an implanted arrhythmia loop recorder
9. Active systemic infection
10. Unstable angina or ongoing myocardial ischemia
11. Myocardial Infarction (MI) within 90 days prior to enrollment
12. Evidence of myxoma, left atrial thrombus or intracardiac mural thrombus++
13. Previous cardiac surgery (i.e. ventriculotomy, atriotomy, CABG, PTCA, PCI, coronary stenting procedures) ≤ 90 days prior to enrollment.
14. Severe valvular disease, including mechanical prosthetic mitral or tricuspid heart valves (patients with successful mitral valve repair allowed - annular ring constitutes repair);
15. Any prior history of documented cerebral infarct, TIA or systemic embolism [excluding a post-operative deep vein thrombosis (DVT)] <180 days prior to enrollment
16. Moderate or severe mitral stenosis (severity assessed on the most recent TTE ≤180 days prior to enrollment. Defined as pulmonary artery systolic pressure >30 mmHg)
17. Presence of left atrial appendage closure device
18. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder
19. Subjects who, in the judgment of the investigator, have a life expectancy of less than two (2) years
20. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon investigator's discretion)
21. Amiodarone use within 60 days prior to enrollment
22. Any carotid stenting or endarterectomy
23. Stage 3B renal disease or higher (estimated glomerular filtration rate, eGFR <45 mL/min)
24. Known coagulopathy disorder (e.g. von Willebrand's disease, hemophilia)
25. Any known contraindication to an AF ablation
26. Any known contraindication for anticoagulation (e.g. patients unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation)
27. Vena cava embolic protection filter devices and/or known femoral thrombus that prevents catheter insertion from the femoral approach
28. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
29. Rheumatic Heart Disease
30. Presence of intramural thrombus, tumor or other abnormality that precludes vascular access, or manipulation of the catheter
31. Subjects unable or unwilling to complete follow-up visits and examinations for the duration of the clinical study
32. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the sponsor to determine eligibility.

    * LVEF and LA diameters obtained ≤180 days prior to enrollment will be acceptable, unless a cardiac event has occurred (e.g. MI) between the date of the exam and the enrollment date. In this case, a new echocardiogram (trans-thoracic or trans-esophageal, or intracardiac echo) must be performed to confirm eligibility prior to performing ablation. If no recent (≤180 days prior to enrollment) echocardiogram is available at the time of the enrollment, a new echocardiogram must be performed either prior to enrolling the patient into the study or post-consent to confirm patient's eligibility prior to performing the ablation. For TTE, LA anteroposterior diameter measured by M-mode from the parasternal long-axis view will be used. If both LA diameter and volume are available and at least one of them meets the exclusion criteria, the subject is considered ineligible for the study.

      * The absence of thrombus must be confirmed by means of a trans-esophageal echocardiogram (TEE) within 48 hours prior to the procedure or Intracardiac Echography (ICE) during the procedure in subjects not adequately anticoagulated per Section 10.4.2. If a thrombus is observed, the subject no longer meets eligibility criteria and should be considered "Consent Ineligible".

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Michaud, Principal Investigator — Massachusetts General Hospital
Locations (47):
- United States (25):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - AdventHealth Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - St. Lukes Idaho Cardiology Associates, Boise, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - St. John's Hospital, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Hospital Medical Center, West Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - Catholic Medical Center, Manchester, New Hampshire
  - Northwell Health, Bay Shore, New York
  - Weill Cornell Medical University, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Bryn Mawr Medical Specialists, Bryn Mawr, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Orion Medical, Pasadena, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Chippenham and Johnston-Willis Hospital (CJW), Richmond, Virginia
- Austria (2):
  - A.o. Krankenhaus der Elisabethinen Linz, Linz
  - Allgemeines Krankenhaus AKH, Vienna
- Onze Lieve Vrouw Ziekenhuis, Aalst, Belgium
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Ste-Foy, Quebec
- Hospital de la Pitie-Salpetriere, Paris, France
- Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau, Germany
- Hong Kong (2):
  - Queen Elizabeth Hospital, Kowloon
  - Prince of Wales Hospital, Shatin
- Italy (2):
  - Az. Osp. Lancisi, Ancona, AN
  - Fondazione Centro San Raffaele, Milan
- Japan (2):
  - Kokura Memorial Hospital, Fukuoka-ken
  - Yokosuka Kyosai Hospital, Kanagawa
- Centre Hospitalier Princesse Grace, Monaco, Monaco
- Medisch Spectrum Twente, Amsterdam, Netherlands
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Papworth Hospital, Cambridge
  - Liverpool Heart and Chest Hospital, Liverpool
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
No request for study data has been made at this time. However, Boston Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 299 subjects were enrolled in the NEwTON AF study and subsequently classified as Treatment subjects undergoing an ablation procedure with the Investigational IntellaNav™ StablePoint Catheter System.
  Of the Treatment subjects, eight (8) were lost to follow-up (2 subjects) or withdrew from the study prior to study completion (6 subjects).
Period: Overall Study
Arm/Group | Treatment With Ablation Catheter
Started | 299
Completed | 291
Not Completed | 8
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Treatment Subjects
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 299
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Enrollment (years)
  years | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 181
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Subjects may contribute to more than one category.
  Participants
    Hispanic or Latino | 5
    Native American | 0
    Asian | 48
    Black | 3
    Pacific Islander | 0
    White | 244
    Other | 1
    Race Undisclosed | 5
Region of Enrollment [Number; unit: participants]
  Hong Kong | 6
  United States | 168
  Japan | 6
  United Kingdom | 13
  Canada | 14
  Austria | 14
  Netherlands | 2
  Belgium | 7
  Monaco | 1
  Taiwan | 33
  Italy | 31
  Germany | 4
Height [Mean (Standard Deviation); unit: cm] — Population: Baseline assessment was completed for 298 of 299 Treatment subjects as baseline was missed for one subject in an oversight.
  cm
    number analyzed (Participants) | 298
    (all) | 172 (11)
Weight [Mean (Standard Deviation); unit: kg] — Population: Baseline assessment was completed for 298 of 299 Treatment subjects as baseline was missed for one subject in an oversight.
  kg
    number analyzed (Participants) | 298
    (all) | 86 (21)
BMI [Mean (Standard Deviation); unit: percentage] — Population: Baseline assessment was completed for 298 of 299 Treatment subjects as baseline was missed for one subject in an oversight.
  percentage
    number analyzed (Participants) | 298
    (all) | 29 (6)
Pulse [Mean (Standard Deviation); unit: bpm] — Population: Baseline assessment was completed for 298 of 299 Treatment subjects as baseline was missed for one subject in an oversight.
  bpm
    number analyzed (Participants) | 298
    (all) | 69 (15)
Systolic BP [Mean (Standard Deviation); unit: mmHg] — Population: Baseline assessment was completed for 298 of 299 Treatment subjects as baseline was missed for one subject in an oversight.
  mmHg
    number analyzed (Participants) | 298
    (all) | 134 (20)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] — Population: Baseline assessment was completed for 298 of 299 Treatment subjects as baseline was missed for one subject in an oversight.
  mmHg
    number analyzed (Participants) | 298
    (all) | 78 (11)
Heart Auscultation [Count of Participants; unit: Participants]
  Normal Heart Sounds | 295
  Other | 4
Baseline 12-lead ECG Rhythm [N (%)] [Count of Participants; unit: Participants]
  Sinus Rhythm | 176
  Sinus Bradycardia | 81
  Atrial Fibrillation (AF) | 29
  Atrial Flutter (Not defined) | 3
  Atrial Flutter (Typical Right Cavo Tricuspid Isthmus dependent) | 1
  Sinus Brady with PAC's | 1
  Ectopic Atrial Bradycardia | 1
  Sinus Rhythm with 1st degree block | 1
  Not Assessed/Reported | 6
Respiratory Rate [Mean (Standard Deviation); unit: breaths per minute] — Population: Baseline measure not calculated for all Treatment subjects.
  breaths per minute
    number analyzed (Participants) | 288
    (all) | 16 (2)
Respiratory Rhythm [Count of Participants; unit: Participants] — Population: Baseline assessment was completed for 298 of 299 Treatment subjects as baseline was missed for one subject in an oversight.
  Participants
    number analyzed (Participants) | 298
    Regular | 296
    Irregular | 2
Lung Auscultation [Count of Participants; unit: Participants]
  Normal | 296
  Crackles | 1
  Rhonchi | 1
  Not Assessed/Reported | 1
Cardiac Disease History [Count of Participants; unit: Participants]
  None | 127
  Ischemic Cardiomyopathy | 1
  Non-ischemic Cardiomyopathy | 8
  Myocardial Infarction | 3
  Angina Pectoris | 12
  Congenital Heart Disease | 1
  Congestive Heart Failure | 16
  Cerebrovascular Disease | 4
  Peripheral Vascular Disease | 8
  Hypertension | 131
  Pulmonary Hypertension | 8
  Dyslipidemia | 93
  Pulmonary Embolism | 4
  DVT | 6
  Other Cardiovascular Disease | 17
Neurological Medical History [Count of Participants; unit: Participants]
  None | 287
  Carotid Artery Disease | 2
  TIA | 7
  CVA | 3
Cardiac Procedure History [Count of Participants; unit: Participants]
  None | 269
  PTCA | 9
  Stent | 15
  CABG | 5
  Pacemaker/ICD/CRT | 0
  Cardiac Valve | 0
  LAAC | 1
  PFO Intervention | 0
  ASD Intervention | 0
  Heart Transplant | 0
  Other Cardiovascular Procedure | 10
Ventricular Arrhythmia History [Count of Participants; unit: Participants]
  None | 264
  Ventricular Tachycardia | 15
  Ventricular Fibrillation | 0
  Other Ventricular Arrhythmia | 25
Atrial Arrhythmia History [Count of Participants; unit: Participants]
  Atrial Fibrillation | 299
  Atrial Tachycardia | 95
  Atrial Flutter | 95
  Typical Atrial Flutter | 73
  Other Atrial Arrhythmia | 18
Brady Arrhythmia History [Count of Participants; unit: Participants]
  None | 183
  Sinus Bradycardia | 107
  Sinus Node Dysfunction | 6
  Sick Sinus Syndrome Chronotropic Incompetence | 4
  Sinus Arrest | 3
  AV Block 1 | 19
  AV Block 2 | 2
  AV Block 3 | 0
  Other Brady Arrhythmia | 1
Cardiac Ablation History [Count of Participants; unit: Participants]
  None | 281
  Any Left Atrial Ablation | 0
  Any Cardiac Ablation | 18
Non-Cardiac Comorbidities [Number; unit: participants]
  None | 147
  COPD | 12
  Diabetes (Type 1) | 2
  Diabetes (Type 2) | 33
  Hepatic Disease | 5
  Renal Disease | 7
  Gastrointestinal Disorder | 42
  Sleep Disordered Breathing | 49
  Other Non-Cardiac Co-Morbidities | 85

OUTCOME MEASURES:

1. Primary Outcome: Rate of Primary Safety Events at 1-Month Post-Procedure
Description: The primary safety endpoint at 30 days is defined as the safety event-free rate at 1-Month (30 days) post-procedure.
Time Frame: Up to 30 Days
Population: Of the 299 treatment subjects, a total of 13 primary safety events occurred through 30 days in 12 subjects.
Measure: Number; unit: primary safety events
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 299
primary safety events | 13

2. Primary Outcome: Rate of Primary Safety Events at 12-Months Post-Procedure
Description: The primary safety endpoint at 12 months is defined as the safety event-free rate at 12 months post-procedure.
Time Frame: 12 Months
Population: Of the 299 treatment subjects, a total of 13 primary safety events occurred through 12 months in 12 subjects.
Measure: Number; unit: primary safety events
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 299
primary safety events | 13

3. Primary Outcome: Percentage of Participants With Freedom From Treatment Failure at 12-Months Post-Procedure
Description: The twelve-month effectiveness endpoint is defined as the event-free rate at twelve-month post-procedure.
Time Frame: 12 Months
Population: The freedom from primary effectiveness failure at 12 months is 60.5%.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 299
Participants | 181

4. Primary Outcome: Number of Participants That Achieved Electrical Isolation of All Pulmonary Veins
Description: The primary effectiveness endpoint of acute procedural success is defined as the achievement of electrical isolation of all PVs using the IntellaNav StablePoint catheter only.
Time Frame: 30 Days
Population: Acute procedural success was observed in 294 (98.3%) of the 299 Treatment subjects that underwent an ablation procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 299
Participants | 294

5. Secondary Outcome: Rate of AEs Through 12-Months Post-Procedure
Description: Secondary Safety Endpoint - AE Rates
Time Frame: 12 Months
Population: Adverse events (AEs) that occurred during the study were continuously monitored. A total of 156 events were reported in 97 of the 299 Treatment subjects.
Measure: Number; unit: Events Reported
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 97
Events Reported | 156

6. Secondary Outcome: Number of Patients With New or Increased Dose of AAD
Description: Secondary Effectiveness Endpoint 1 - New or Increased Dose of AAD
Time Frame: 12 Months
Population: Subjects were only counted as effectiveness failures if a new AAD or higher dose of a previously failed AAD continued after the blanking period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 296
Participants
  Subjects with New or Increased Dose of AAD | 103
  Subjects with No New or Increased Dose of AAD | 193

7. Secondary Outcome: Percentage of Participants With Freedom From Primary Effectiveness Failure Without a Repeat Procedure
Description: Secondary Effectiveness Endpoint 2 - Single Procedure Success defined as freedom from primary effectiveness failure without a repeat procedure
Time Frame: 12 Months
Population: 59% of subjects were free from primary effectiveness failure without a repeat procedure at 12-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 296
Participants | 175

8. Secondary Outcome: Percentage of Participants With Freedom From Documented Symptomatic Atrial Fibrillation, Atrial Flutter and Atrial Tachycardia Recurrence
Description: Secondary Effectiveness Endpoint 3 - Symptomatic Recurrence: freedom from documented symptomatic AF/AT/AFL recurrence
Time Frame: 12 Months
Population: The freedom from documented arrhythmia recurrence, including atrial fibrillation (AF), atrial flutter (AFL), and atrial tachycardia (AT), was 71%.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 294
Participants | 211

9. Secondary Outcome: Rate of SAEs Through 12-Months Post-Procedure
Description: Secondary Safety Endpoint - SAEs
Time Frame: 12 Months
Population: Adverse events (AEs) that occurred during the study were continuously monitored. A total of 156 events were reported in 97 of the 299 Treatment subjects. A total of 72 Serious Adverse Events (SAEs) were reported in 47 Treatment subjects.
Measure: Number; unit: Total number of reported SAEs
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 47
Total number of reported SAEs | 72

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment With Ablation Catheter
All-Cause Mortality (participants affected / at risk) | 0/299
Serious Adverse Events (participants affected / at risk) | 47/299
Other Adverse Events (participants affected / at risk) | 64/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Ablation Catheter (N=299)
Atrial flutter, not specified (Surgical and medical procedures) | 1 (1) — Ablation Related
Fistula (Arterial/Venous) (Surgical and medical procedures) | 1 (1) — Ablation Related
Hemodynamic Instability (Surgical and medical procedures) | 1 (1) — Ablation Related
Myocardial Perforation with Tamponade (Surgical and medical procedures) | 1 (1) — Ablation Related
Oozing/Bleeding (Surgical and medical procedures) | 1 (1) — Ablation Related
Pericardial Effusion (Surgical and medical procedures) | 3 (3) — Ablation Related
Pericarditis (Surgical and medical procedures) | 6 (6) — Ablation Related
Post procedure infection/sepsis (Surgical and medical procedures) | 1 (1) — Ablation Related
Procedure related Abnormal labs (Surgical and medical procedures) | 1 (1) — Ablation Related
Procedure related Allergic reactions/Adverse drug reaction (Surgical and medical procedures) | 1 (1) — Ablation Related
Procedure related anesthesia/sedation (Surgical and medical procedures) | 2 (2) — Ablation Related
Procedure related Gastrointestinal (Surgical and medical procedures) | 2 (2) — Ablation Related
Procedure related Genitourinary/Renal (Surgical and medical procedures) | 1 (1) — Ablation Related
Pseudoaneurysm (Surgical and medical procedures) | 1 (1) — Ablation Related
Pulmonary Thromboembolism (Surgical and medical procedures) | 1 (1) — Ablation Related
Pulmonary Edema (Surgical and medical procedures) | 2 (2) — Ablation Related
Right atrial (Type I) atrial flutter (Surgical and medical procedures) | 1 (1) — Ablation Related
Sinus bradycardia (Surgical and medical procedures) | 1 (1) — Ablation Related
Stroke (Surgical and medical procedures) | 1 (1) — Ablation Related
Atrial Fibrillation (AF) (Cardiac disorders) | 4 (4) — Cardiovascular
Atrial Flutter (Cardiac disorders) | 2 (2) — Cardiovascular
Atrial tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 1 (2) — Cardiovascular
Coronary artery disease (Cardiac disorders) | 2 (2) — Cardiovascular
Dyspnea - Heart Failure (Cardiac disorders) | 1 (1) — Cardiovascular
Heart Failure symptoms - Unspecified (Cardiac disorders) | 1 (1) — Cardiovascular
Infection - Unrelated procedure/device (Cardiac disorders) | 1 (1) — Cardiovascular
Multiple Symptoms (Cardiac disorders) | 1 (1) — Cardiovascular
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 1 (1) — Cardiovascular
Abnormal laboratory values (General disorders) | 2 (2) — Non-Cardiovascular
Adverse reaction - Medication (General disorders) | 1 (1) — Non-Cardiovascular
Cancer (General disorders) | 2 (2) — Non-Cardiovascular
Fever and/or virus (General disorders) | 2 (2) — Non-Cardiovascular
Gastrointestinal (General disorders) | 3 (5) — Non-Cardiovascular
Head, Eyes, Ears, Nose, Throat (HEENT) (General disorders) | 1 (1) — Non-Cardiovascular
Hematological (General disorders) | 2 (3) — Non-Cardiovascular
Musculoskeletal (General disorders) | 4 (4) — Non-Cardiovascular
Neurological (General disorders) | 2 (2) — Non-Cardiovascular
Physical Trauma (General disorders) | 1 (1) — Non-Cardiovascular
Psychological (General disorders) | 1 (1) — Non-Cardiovascular
Pulmonary (General disorders) | 4 (4) — Non-Cardiovascular
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Ablation Catheter (N=299)
Angina/Chest pain (Surgical and medical procedures) | 1 (1) — Ablation Related
Atrial Fibrillation (AF) (Surgical and medical procedures) | 2 (2) — Ablation Relate
Atrial flutter, not specified (Surgical and medical procedures) | 1 (1) — Ablation Related
Bleeding related to anticoagulation (Surgical and medical procedures) | 1 (1) — Ablation Related
Edema (Surgical and medical procedures) | 1 (1) — Ablation Related
Hematoma (Surgical and medical procedures) | 2 (2) — Ablation Related
Nerve Damage (Surgical and medical procedures) | 1 (1) — Ablation Related
Oozing/Bleeding (Surgical and medical procedures) | 3 (3) — Ablation Related
Pain (Non-cardiovascular) (Surgical and medical procedures) | 3 (3) — Ablation Related
Pain cardiovascular (Non-ischemic) (Surgical and medical procedures) | 3 (3) — Ablation Related
Pericardial effusion (Surgical and medical procedures) | 2 (2) — Ablation Related
Pericarditis (Surgical and medical procedures) | 16 (16) — Ablation Related
Pleuritis (Surgical and medical procedures) | 1 (1) — Ablation Related
Post procedure infection/sepsis (Surgical and medical procedures) | 3 (3) — Ablation Related
Post procedure wound discomfort (Surgical and medical procedures) | 1 (1) — Ablation Related
Procedure related Allergic reactions/Adverse drug reaction (Surgical and medical procedures) | 2 (2) — Ablation Related
Procedure related Anesthesia/Sedation (Surgical and medical procedures) | 3 (3) — Ablation Related
Procedure related Gastrointestinal (Surgical and medical procedures) | 1 (1) — Ablation Related
Procedure related Genitourinary/Renal (Surgical and medical procedures) | 4 (4) — Ablation Related
Procedure related Hypertension (Surgical and medical procedures) | 1 (1) — Ablation Related
Procedure related Neurological (Non-TIA, non-stroke, dysphagia, speech disturbance/dysarthria) (Surgical and medical procedures) | 1 (1) — Ablation Related
Procedure related Pulmonary (including cough, hemoptysis) (Surgical and medical procedures) | 1 (1) — Ablation Related
Stroke (Surgical and medical procedures) | 1 (1) — Ablation Related
Visual blurring/disturbances (Surgical and medical procedures) | 2 (2) — Ablation Related
Atrial Fibrillation (AF) (Cardiac disorders) | 7 (8) — Cardiovascular
Atrial flutter (Cardiac disorders) | 1 (1) — Cardiovascular
Chest pain - Other (Cardiac disorders) | 2 (2) — Cardiovascular
Distal thromboemboli (Cardiac disorders) | 1 (1) — Cardiovascular
Multiple Heart Failure symptoms (Cardiac disorders) | 1 (1) — Cardiovascular
Multiple symptoms (Cardiac disorders) | 1 (1) — Cardiovascular
Palpitations (Cardiac disorders) | 1 (1) — Cardiovascular
Sinus bradycardia (Cardiac disorders) | 1 (1) — Cardiovascular
Adverse reaction - Medication (General disorders) | 1 (1) — Non-Cardiovascular
Fever and/or virus (General disorders) | 5 (5) — Non-Cardiovascular
Gastrointestinal (General disorders) | 1 (1) — Non-Cardiovascular
Genitourinary (General disorders) | 2 (2) — Non-Cardiovascular
Hematological (General disorders) | 1 (1) — Non-Cardiovascular
Neurological (General disorders) | 1 (1) — Non-Cardiovascular

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT04580914/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04580914/ICF_001.pdf